CLINICAL TRIAL: NCT06932965
Title: Assessment of the Effects of Cervical Stabilization Exercises and Proprioception Training on Balance and Posture in Individuals With Forward Head Posture
Brief Title: Cervical Exercises and Balance in Forward Head Posture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nevsehir Haci Bektas Veli University (Other)
Responsible Party: Principal Investigator, Muhammet Ozalp, Assistant Professor, PhD, Physiotherapist, Nevsehir Haci Bektas Veli University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NevsehirHBVUKozakli
Record Dates: First submitted 2025-04-10; First posted 2025-04-17 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Forward Head Posture
Keywords: cervical stabilization; proprioception; forward head posture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control (No Intervention): no intervention only measurement
- Cervical Stabilization Group (Experimental): Participants performed supervised cervical stabilization exercises for 8 weeks, 3 sessions per week.
  Interventions: Behavioral: Cervical Stabilization Group
- Combined Group (Experimental): Participants performed both exercise protocols as described above over the same period.
  Interventions: Behavioral: combined group

INTERVENTIONS:
Behavioral: Cervical Stabilization Group — Participants performed supervised cervical stabilization exercises for 8 weeks, 3 sessions per week.
  Arms: Cervical Stabilization Group
Behavioral: combined group — Participants performed both exercise protocols as described above over the same period
  Arms: Combined Group

SUMMARY:
This study aims to evaluate the effects of neck stabilization exercises and proprioception training on balance and posture in university students aged 18-25 who are detected to have forward head posture.

Individuals will be evaluated before the study, and following the evaluation, stabilization exercises will be applied to the first group under the control of a physiotherapist 3 days a week for 6 weeks. In addition to the stabilization exercises, proprioception training will be given to the second group. Individuals are trained with cervical proprioceptive training, exercises performed by returning the neck to its natural neutral posture and to positions within a predetermined range.

Patients are first trained with their eyes open, then with their eyes closed. Feedback for proprioceptive performance is necessary to reduce the margin of error in repositioning. Laser pointer headbands were used for feedback. With the help of this laser pointer, exercises will be applied to the patients by increasing the level of difficulty. In order to make the exercises more difficult, they will first be applied sitting, then standing, then in semi-tandem and tandem positions. No program will be applied to the 3rd group, the control group.

DETAILED DESCRIPTION:
This study aims to evaluate the effects of neck stabilization exercises and proprioception training on balance and posture in university students aged 18-25 who were found to have forward head posture.

This study was designed with a randomized controlled experimental research model. Following the ethics committee approval, the data of the study will be collected in the Nevşehir Hacı Bektaş Veli University Kozakli Vocational School Application Laboratory.

Inclusion Criteria for the Study:

University students aged 18-25, Those with a craniovertebral angle (CVA) less than 50 degrees, (34). No history of trauma or surgery in the neck region, No systemic disease, No dizziness problems, Individuals who want to participate in the study voluntarily, Individuals who have received informed consent

Exclusion criteria:

Patients who are not between the ages of 18-25, those with a craniovertebral angle greater than 50 degrees, those who are mentally incapable of making assessments, those who cannot adapt to the training program and those who refuse to participate in the study will not be included.

Individuals will be evaluated before the study, following the evaluation, stabilization exercises will be applied to the first group 3 days a week for 6 weeks under the control of a physiotherapist. In addition to the stabilization exercises, the second group will receive proprioception training. Individuals are trained with cervical proprioceptive training, exercises performed by returning the neck to its natural neutral posture and to positions within a predetermined range.

Patients are first trained with their eyes open, then with their eyes closed. Feedback for proprioceptive performance is necessary to reduce the margin of error in repositioning. Laser pointer headbands were used for feedback. With the help of this laser pointer, exercises will be applied to the patients by increasing the level of difficulty. In order to make the exercises more difficult, they will first be applied sitting, then standing, then in semi-tandem and tandem positions. No program will be applied to the 3rd group, the control group.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged between 18-35
* Diagnosed with forward head posture based on craniovertebral angle
* No prior neck surgery or trauma
* Able to participate in exercise sessions

Exclusion Criteria:

* Neurological or musculoskeletal disorders affecting balance
* Recent injury or surgery in cervical spine
* Use of medications affecting postural control

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
CVA | baseline
  Participants were included when they have a CVA < 54°, had no cervical trauma or surgical history, systemic disease, and dizziness problem. We fixed the camera (Nikon D5100) 1.5 meters away from the individual and at the shoulder level. According to radiography, which is considered the gold standard in determining the head forward posture, measurements made by photography were found to be valid and reliable (Van Niekerk et al., 2008). A self-balanced position was chosen and side-shots were taken. The examiner marked the C7 spinous process as well as the tragus of the ear. The CVA is calculated at the intersection angle of a line extending to the ear's tragus and a horizontal line passing the spinous of C7. We used Adobe Acrobat software to measure the angle. CVA less than 54 is defined as FHP. We did not include the individual in the study if the CVA was 54 degrees or greater
Y-Balance Test (YBT) | baseline and after 8 weeks
  This test, an adaptation of the Star Excursion Balance Test (SEBT), was employed to assess the dynamic balance of participants. This evaluation was conducted for both feet, starting with the dominant leg positioned at the center of the test. Three reaching directions-anterior, posteromedial, and posterolateral-were incorporated into the test, with the apparatus pulled using three tape measures between 90° and 135° in these directions. Participants were instructed to reach as far as possible along the specified line, touching the ground with the most distal part of the reaching foot. Subsequently, they were required to return the reaching leg to a double-leg stance while maintaining a single-leg stance. The test was performed clockwise or counterclockwise, corresponding to the dominance of the right or left leg, respectively. Participants were instructed to keep their hands on the iliac crest and ensure that the heels of the standing legs remained in contact with the ground throughout.

SECONDARY OUTCOMES:
Joint Position Sense | Baseline and after 8 weeks
  Cervical proprioceptive evaluation was based on the evaluation method used by Revel et al. (1991) (4, 27, 28). Participants were asked to sit relaxed on the experimental chair while putting hands on their legs and keeping heads and necks in a self balanced position. Rubbery headbands were prepared, which can be flexibly fixed to the heads of individuals. The laser marker was fixed on top of these headbands. To determine the neutral position's error deviations, a wall was placed 90 cm in front of the individual, parallel to the 1 mm x 1 m sized millimetric papers. Individuals were tested 10 times in each direction, with the eyes open. In the test, we said that the subjects should be in the posture of rest where they feel comfortable. After the cervical flexure's maximal movement from the subjects, they were asked to return their head to a self-balanced position, where they felt their head straight. When they found a neutral position (0 point), they were asked to concentrate on this pos
Stork Balance Test | Baseline and after 8 weeks
  The participant was positioned in a comfortable stance, standing on both feet with hands placed on the hips. They were instructed to lift one leg and place the toes against the knee of the other leg. Following this, the participant was directed to raise the heel and stand on their toes upon command. The stopwatch was initiated as the heel left the floor and stopped under various conditions: if the hand(s) disengaged from the hips, if the supporting foot swiveled or moved in any direction, if the non-supporting foot lost contact with the knee, or if the heel of the supporting foot touched the floor . Each participant underwent three attempts for the test, and the average of these attempts was recorded.
Postural Assessment | Baseline and after 8 weeks
  Measured via photogrammetry for craniovertebral angle.
Balance Performance | Baseline and after 8 weeks
  stork an y-balance test

CONTACTS AND LOCATIONS:
Locations (1):
- Kozakli Vocational School, Nevşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data (IPD).

REFERENCES:
- [Derived] Ozalp M, Talu B, Kayabinar E. Assessment of the effects of cervical stabilization exercises and proprioception training on balance and posture in individuals with forward head posture. BMC Musculoskelet Disord. 2025 Nov 21;26(1):1077. doi: 10.1186/s12891-025-09259-7. PMID 41272563